CLINICAL TRIAL: NCT05141045
Title: The Effect of Fish Oil Supplementation on Vocal Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1708288-3
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Voice Range Profile; Reflux Symptom Index; Evaluation of Ability to Sing Easily; Body Composition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 PUFA supplement (Experimental): omega-3 PUFA supplement, 3.0 grams per day
  Interventions: Dietary Supplement: omega-3 PUFA supplement
- placebo (Placebo Comparator): safflower oil, 3.0 grams per day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 PUFA supplement — participants were instructed to take 3.0 grams per day of omega-3 PUFA supplement
  Arms: omega-3 PUFA supplement
Dietary Supplement: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study was to determine if use of omega-3 PUFA supplement in combination with a singer's training regimen enhances training adaptations and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy college vocal performers (male and female of all ethnicities) *Between the ages of 18-28 years
* Majoring in classical voice in the Baylor University School of Music or musical theatre in the Baylor University Department of Theatre Arts.

Exclusion Criteria:

* Previously diagnosed with a voice disorder
* Vegans
* Smokers
* Allergic to fish, shellfish or safflower oil
* Have been taking daily FO n-3 supplement within the past three months, or any supplement known to effect muscle biology (e.g. creatine).

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Change in Evaluation of Ability to Sing Easily | baseline and up to 11 weeks
  survey designed to aid in subject self-assessment

SECONDARY OUTCOMES:
change in Voice Range Profile | baseline and up to 11 weeks
  known as a phonetogram, is a representation of a participants minimum and maximum intensity levels across vocal range
change in Body composition | baseline and up to 11 weeks
  height in cm, weight measured in kg. Bio-electrical impedance scale use to assess lean and body fat mass, measured in kg. Weight and height were combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: LesLee Funderburk, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No